CLINICAL TRIAL: NCT03430518
Title: A Phase Ib Study Evaluating the Safety and Tolerability of Durvalumab (MEDI4736) (Anti-PDL1) in Combination With Eribulin in Patients With HER2-Negative Metastatic Breast Cancer and Recurrent Ovarian Cancer
Brief Title: Durvalumab and Eribulin in Her2-negative Metastatic Breast Cancer and Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amy Tiersten (Other)
Collaborators: AstraZeneca (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor-Investigator, Amy Tiersten, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-2320
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: HER2-Negative Metastatic Breast Cancer; Recurrent Ovarian Cancer
Keywords: Durvalumab (MEDI4736) (Anti-PDL1); Eribulin; Recurrent Ovarian cancer; Her2-negative Metastatic Breast Cancer; Ovarian cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — durvalumab; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Her2-negative Metastatic Breast Ca and Recurrent Ovarian Ca (Experimental): Durvalumab and Eribulin in Her2-negative Metastatic Breast Cancer and Recurrent Ovarian cancer
  Interventions: Drug: Durvalumab; Drug: Eribulin

INTERVENTIONS:
Drug: Durvalumab — 1.12g given IV on day 1 every 21 day cycle
Drug: Eribulin — 1.1 mg/m2 IV on day 8 of every 21 day cycle in the first 3 patients, then increased to 1.4mg/m2 IV on day 1 and day 8 of every 21 day cycle. If significant toxicity occurs in patients given the 1.1mg/m2 IV dose, then subsequent patients with receive eribulin 0.7mg/m2 IV on day 1 and day 8 of every 21 day cycle.

SUMMARY:
This study will evaluate the recommended Phase 2 combination dose (RP2D) of eribulin with durvalumab.

DETAILED DESCRIPTION:
STUDY SUMMARY

Study Duration: Accrual will take place over the course of 16 months. Patients will be treated until unacceptable toxicity or disease progression (expected on average for 6 months) and then followed for one year thereafter.

Objectives: Phase I: To determine the the recommended phase II dose of eribulin in combination with Durvalumab

This study will evaluate the recommended Phase 2 combination dose (RP2D) of eribulin with durvalumab. If two or more out of 6 patients experience a dose limiting toxicity (DLT) at dose level I or II, the dose level below that level will be considered the RP2D. If all 3 patients enter dose level-I and experience DLT, the study will be terminated. If the highest level has been reached and < 33% of patients have experienced DLT, that will be considered the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization obtained from the subject and documented according to local regulatory requirements prior to beginning any protocol-specific procedures, including screening procedures
* The subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations, including all follow-up
* The subject is medically fit for protocol therapy and competent to give informed consent
* The subject must have a performance status of 0-1 as determined by criteria set forward by ECOG
* Subjects with histologically confirmed stage IV any hormone receptor (HR) status/HER2 negative breast cancer or advanced/recurrent epithelial ovarian cancer

  * HR positive, HER2 negative breast cancer: patients must have received at least one line of therapy for metastatic disease prior to enrollment, including hormonal therapy and a CDK4/6 inhibitor
  * HR negative, HER2 negative breast cancer: patients must have received at least one prior line of chemotherapy for metastatic disease
  * Recurrent, "platinum-sensitive" epithelial ovarian cancer: patients must have received at least two lines of platinum-based chemotherapy prior to enrollment, with at least one of these lines of platinum-based chemotherapy in the recurrent setting
  * Recurrent, "platinum-resistant" (recurrence within 6 months of a platinum-containing chemotherapy regimen) epithelial ovarian cancer: patients must have received at least one line of platinum-based chemotherapy prior to enrollment
* There is pathologic tissue confirming of metastatic breast or ovarian cancer
* All adverse events from prior chemotherapy, radiation, or surgery have either returned to baseline or are < grade 1 prior to administration of the investigational product
* The subject has a body weight of greater than 30kg
* The subject must have at the time of screening acceptable hematologic, hepatic, and renal function, defined by the following (≤ 28 days prior to registration):
* Absolute neutrophil count > 1500/mm3
* Hemoglobin > 10g/dL
* Platelet count > 100,000/mm3
* Creatinine < 1.6 mg/dL
* Serum creatinine clearance >40mL/min by the Cockcroft-Gault formula or by 24-hour urine collection
* Serum bilirubin < 1.5x the upper limit of institutional normal, excluding patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology)
* Transaminases (AST/SGOT and ALT/SGPT) < 2.5 times above the upper limits of the institutional normal, unless liver metastases are present, in which case it must be < 5x ULN
* INR < 2 for patients who are not on systemic anticoagulation. Patients on anticoagulation therapy with an INR > 2 may be enrolled at the discretion of the investigator if they have not had any episodes of severe hemorrhage or active bleeding
* The subject must be 18 years of age or older
* The subject must have not had more than 5 prior lines of cytotoxic chemotherapy in the metastatic setting, not including hormonal therapies
* Evidence of post-menopausal status, history of hysterectomy or bilateral oophorectomy, or negative serum or urine pregnancy test within 7 days prior to starting treatment

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have LH and FSH levels in the post-menopausal range for the institution
  * Women > 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, or had chemotherapy-induced menopause with last menses >1 year ago
* Women of child-bearing potential must agree to use at least one highly effective form of contraception beginning at least 28 days prior to study entry, continuing to do so for the duration of their participation in the study, and for 90 days after the last dose of study drug. Non-sterilized male partners must also agree to use a male condom plus spermicide for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of childbearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months without alternative medical cause), as defined above in section 3.1.1

Exclusion Criteria:

* Prior treatment with any investigational drug as part of a clinical trial within 28 days prior to study drug administration
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* The subject has been treated previously with any anti-PD1/PDL1 therapy, including durvalumab
* The subject has been previously treated with eribulin
* The subject has received a prior anti-cancer therapy (chemotherapy, targeted small molecule therapy, endocrine therapy, immunotherapy, biologic therapy, tumor embolization, monoclonal antibodies) within 14 days prior to study Day 1
* Any concurrent anti-cancer therapy other than denosumab, bisphosphonates, or hormonal therapy for non-cancer related conditions
* The subject has received radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 28 days of the first dose of study drug
* Major surgical procedure within 28 days prior to the first dose of study drug (local surgery or isolated lesions for palliative intent is acceptable)
* Any unresolved toxicity NCI CTCAE Grade >2 from previous anticancer therapy with the exception of alopecia, vitiligo, and lab values which meet inclusion criteria

  * Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study as per consultation with the study physician. These patients will require active and continuous monitoring of this toxicity and if any worsening is observed or identified, study drugs will be permanently discontinued immediately
  * Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with eribulin or durvalumab may be included after consultation with the study physician
* The subject has a history of, or is reasonably suspected to meet criteria for the diagnosis of a known congenital or acquired disorder causing systemic immunosuppression or immunodeficiency
* The subject has a history of allogeneic organ or bone marrow transplantation
* The subject has a history of, or is reasonably suspected to meet criteria for the diagnosis of a systemic auto-immune/inflammatory disease or other autoimmune disorder, including but not limited to inflammatory bowel disease (Crohn's disease or ulcerative colitis), active diverticulitis, systemic lupus erythematosus, Sarcoidosis, Wegener's granulomatosis, granulomatosis with polyangiitis, pneumonitis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis.

  * Exceptions: vitiligo, alopecia, autoimmune-related hypothyroidism which is stable on hormone replacement, chronic skin conditions that do not require systemic therapy, celiac disease controlled with diet alone, or any subjects without active disease in the last 5 years if deemed appropriate by the study physician
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exception of inhaled, local injection, or intranasal corticosteroids, systemic steroids at physiological doses (equivalent of ≤ 10mg prednisone daily), and steroid premedication for hypersensitivity reactions (e.g., CT scan premedication)
* The subject has known active central nervous system (CNS) metastases, spinal cord compression, and/or leptomeningeal carcinomatosis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. Following radiotherapy and/or surgery for brain metastases subjects must wait 4 weeks following the intervention before enrollment to confirm stability.
* The subject has a current or past history of active TB (Bacillus Tuberculosis)
* The subject has an active infection requiring systemic therapy
* The subject has HIV disease (positive HIV 1/2 antibodies)
* The subject has active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] PCR is detected). Subjects with a past or resolved HBV infection (HBcAb positive and absence of HBsAg reactivity) are eligible
* The subject has received a live virus vaccine within 30 days of planned start of study therapy Note: Seasonal influenza vaccines for injection are generally inactivated. Flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* The subject has a known additional malignancy that is progressing or requires active treatment. Exceptions include non-melanoma cancers of the skin that have been resected, in situ malignancies that have been managed with curative therapy and there is no current evidence of disease at time of trial enrollment, or history of prior malignancy with no known active disease for 5 years prior to trial enrollment
* Female patients who are pregnant or breast feeding
* Subject is of reproductive potential and is not willing to use effective birth control methods from screening for 90 days after the last dose of durvalumab
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab or eribulin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study including but not limited to:

  * Symptomatic congestive heart failure of New York Heart Association Class III or IV
  * Mean QT interval corrected for heart rate (QTc) > 470ms calculated from 3 electrocardiograms within 15 minutes at 5 minutes apart using Fridericia's Correction
  * Unstable angina pectoris, uncontrolled hypertension, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Interstitial lung disease, or severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 89% or less at rest on room air
  * Serious chronic gastrointestinal conditions associated with diarrhea
  * A known or active bleeding diathesis
  * Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial or increase risk of adverse events
  * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
  * Active (acute or chronic) or uncontrolled infections
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
The dose-limiting toxicity (DLT) rate | 42 days
  A DLT is defined as a ≥ Grade 3 or 4 study drug-related adverse event (using NCI CTCAE Version 4.03) that occurs during the DLT evaluation period. Toxicity that is clearly and directly related to the primary disease or to another etiology is excluded from this definition.

SECONDARY OUTCOMES:
Number of Adverse events | 6 months
  Adverse events associated with eribulin when administered in combination with durvalumab will be described according to the Medical Dictionary for Regulatory Activities (MedDRA) by system organ classes.
Objective response rate (ORR) | 6 months
  Objective response rate (ORR) is measured as the proportion of patients who have achieved complete response, partial response (CR, PR) according to Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria. irCR, complete disappearance of all measurable and non-measurable lesions. Lymph nodes must decrease to < 10 mm in short axis. Confirmation of response is not mandatory. irPR, decrease of ≥ 30% in TMTB relative to baseline, non-target lesions are irNN, and no unequivocal progression of new non-measurable lesions.
Progression free survival (PFS) | 16 months
  Progression free survival (PFS) is measured from the start of first treatment until the criteria for progression are met or death, whichever occurs earlier. Patients without documented progression/death will be censored at the last disease assessment date.
Overall survival (OS) | 6 months
  Overall survival (OS) is measured from the start of first treatment until death due to any cause. Patients without documented death at the time of analysis will be censored at the date last known to be alive.
ECOG performance status | 6 months
  Eastern Cooperative Oncology Group (ECOG) performance status. Grade 0: Fully active, able to carry on all pre-disease performance without restriction Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours Grade 4: Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair Grade 5: Dead

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No